CLINICAL TRIAL: NCT04692116
Title: EarlyFocus I: A Single Center Study on the Short-term Safety of Parkinson's Disease (PD) Treated With Focused Ultrasound Subthalamotomy at an Early Stage (<5 Years From the Diagnosis).
Brief Title: Parkinson's Disease (PD) Treated With Focused Ultrasound Subthalamotomy at an Early Stage
Acronym: EarlyFocus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Collaborators: Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD020
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single-site open clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExAblate Arm (Experimental): ExAblate Model 4000 System for the treatment of Parkinson's disease
  Interventions: Device: ExAblate treatment

INTERVENTIONS:
Device: ExAblate treatment — Subthalamotomy using the ExAblate

SUMMARY:
Parkinson's disease (PD) is a common, progressive, incurable neurodegenerative disease that can result in severe disability and impairment in health-related quality of life. Current medical and surgical therapies are aimed toward maximal symptom relief with minimal associated side effects or morbidity. It is generally accepted that a well-placed stereotactic lesion is comparable in its magnitude of clinical effect to the high frequency electrical stimulation of the same target.

Exablate Neuro is intended to treat movement disorders with unilateral ablation of targets in the thalamus, subthalamic nucleus and globus pallidus nuclei.

With the ExAblate system, transcranial high-intensity focused ultrasound has been coupled with high resolution MRI to provide precise, consistent treatments that can be monitored throughout the procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-65 years old.
2. Subjects who are able and willing to give consent and able to attend all study visits.
3. Diagnosis of PD according to UK (United Kingdom) Brain Bank Criteria as confirmed by movement disorder neurologist at our centre.
4. Less than 5 years since first PD diagnosis.
5. F-dopa PET (Positron Emission Tomography) pattern of striatal dopaminergic denervation suggestive of Parkinson's disease (rostro-caudal gradient).
6. Stable pharmacological regime for the 4-weeks prior to procedure.
7. Topographic coordinates of the subthalamic nucleus are localizable on MRI (Magentic Resonance Imaging) so that it can be targeted by the ExAblate device.
8. Able to communicate sensations during the ExAblate MRgFUS treatment.

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2.5 or greater
2. Presence of severe dyskinesia as noted by a score of 3 or 4 on questions 4.1 and 4.2 of the MDS-UPDRS.
3. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
4. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
5. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
6. Presence of significant cognitive impairment defined as score ≤ 21 on the Montreal Cognitive Assessment (MoCA) or Mattis Dementia Rating Scale of 120 or lower.
7. Patients without clinically relevant parkinsonism in the off-state as evaluated by two examining neurologists. (or MDS-UPDRS in the most affected side <10).
8. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
9. Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory.
10. Legal incapacity or limited legal capacity as determined by the neuropsychologist
11. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within the preceding 12-month period:

    * Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
    * Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
    * Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
    * Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
12. Subjects with unstable cardiac status including:

    * Unstable angina pectoris on medication
    * Subjects with documented myocardial infarction within six months of protocol entry
    * Significant congestive heart failure defined with ejection fraction < 40
    * Subjects with unstable ventricular arrhythmias
    * Subjects with atrial arrhythmias that are not rate-controlled
13. Severe hypertension (diastolic BP > 100 on medication).
14. History of or current medical condition resulting in abnormal bleeding and/or coagulopathy.
15. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
16. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
17. Patient with severely impaired renal function with estimated glomerular filtration rate <30mL/min/1.73m 2 (or per local standards should that be more restrictive) and/or who is on dialysis;
18. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
19. Significant claustrophobia that cannot be managed with mild medication.
20. Subject who weight more than the upper weight limit of the MR table and who cannot fit into the MR scanner
21. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
22. History of intracranial hemorrhage
23. History of multiple strokes, or a stroke within past 6 months
24. Subjects with a history of seizures within the past year
25. Subjects with malignant brain tumors
26. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
27. Any illness that in the investigator's opinion preclude participation in this study.
28. Subjects unable to communicate with the investigator and staff.
29. Pregnancy or lactation.
30. Subjects who have an Overall Skull Density Ratio lower than 0.42 as calculated from the screening CT.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) associated with ExAblate | Month 6 after the subthalamotomy
  Incidence of Adverse Events (AEs) associated with ExAblate
Severity of Adverse Events (AEs) associated with ExAblate | Month 6 after the subthalamotomy
  Severity of Adverse Events (AEs) associated with ExAblate

SECONDARY OUTCOMES:
Mean change in the motor MDS-UPDRS | Month 3 and 6 after the subthalamotomy
  Mean change in the motor MDS-UPDRS (Movement Disorder Scale-Unified Parkinson's Disease Rating Scale) score in both off- and on-medication conditions (when applicable) for both the treated body side and the total motor score.
  [Lowest score = 0; Highest score = 52; Best outcome = lower score]
Mean change in specific PD motor features | Month 3 and 6 after the subthalamotomy
  Mean change in specific PD motor features of the treated body side (i.e., tremor, rigidity and akinesia according to MDS-UPDRS III subscores [Movement Disorder Scale-Unified Parkinson's Disease Rating Scale III].
MDS-UPDRS I score [Movement Disorder Scale-Unified Parkinson's Disease Rating Scale I] | Month 3 and 6 after the subthalamotomy
  Lowest score = 0; Highest score = 52; Best outcome = lower score
MDS-UPDRS II score [Movement Disorder Scale-Unified Parkinson's Disease Rating Scale II] | Month 3 and 6 after the subthalamotomy
  Lowest score = 0; Highest score = 52; Best outcome = lower score
UPDRS IV score [Unified Parkinson's Disease Rating Scale IV] | Month 3 and 6 after the subthalamotomy
  Lowest score = 0; Highest score = 24; Best outcome = lower score
MDS-Non motor rating scale [Movement Disorder Scale] | Month 3 and 6 after the subthalamotomy
  Lowest score = 0; Highest score = 52; Best outcome = lower score
Quality of life assessment (QoL) | Month 3 and 6 after the subthalamotomy
  Assessment of QoL by using the instrument PDQ39
Levodopa equivalent dose change usage | Month 3 and 6 after the subthalamotomy
  Levodopa equivalent dose change usage (milligrams) when applicable

CONTACTS AND LOCATIONS:
Overall Officials: José Obeso, MD, Principal Investigator — Director
Locations (1):
- Hospital Universitario HM Puerta del Sur, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez Fernandez R, Natera Villalba E, Rodriguez-Rojas R, Del Alamo M, Pineda-Pardo JA, Obeso I, Mata-Marin D, Guida P, Jimenez-Castellanos T, Perez-Bueno D, Duque A, Manez Miro JU, Gasca-Salas C, Matarazzo M, Obeso JA. Unilateral focused ultrasound subthalamotomy in early Parkinson's disease: a pilot study. J Neurol Neurosurg Psychiatry. 2024 Feb 14;95(3):206-213. doi: 10.1136/jnnp-2023-331211. PMID 37673642